CLINICAL TRIAL: NCT02285296
Title: The Needs and Burden of Family Caregivers of Older Adults With Cancer and Their Social Determinants
Brief Title: The Needs and Burden of Family Caregivers of Older Adults With Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment problem
Sponsor: University Hospital, Lille (Other)
Collaborators: Centre Oscar Lambret (Other); University of Lille Nord de France (Other); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013_40; 2014-A00018-39 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Oncologic Disorders; Tumor
Keywords: geriatric assessment; Caregivers; Needs Assessment; oncology nursing; frail elderly; Medical, psychologic and sociologic approach
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control arm (No Intervention): usual care
- personalized support program (Experimental): interview of the primary caregivers to identify their needs and expectations, the implementation of a "personalized support program", including telephone follow-up
  Interventions: Other: personalized support program

INTERVENTIONS:
Other: personalized support program — interview of the primary caregivers to identify their needs and expectations, the implementation of a "personalized support program", including telephone follow-up
  Arms: personalized support program

SUMMARY:
Elderly cancer patients need more help from their relatives and for longer than young adults.

Our hypothesis of research is that the needs and resources to help the couple " elderly patient/caregiver ", are at least in part socially determined and that the implementation of a personalized support plan to help the caregiver (PSP) taking into account needs, resources and expectations of the primary caregiver in addition to those of elderly patients with cancer may partly correct inequalities. The PSP should allow a better management of cancer, a lesser burden for the caregiver and a better quality of life for both the caregiver and the patient.

DETAILED DESCRIPTION:
Scientific context Elderly cancer patients need more help from their relatives and for longer than young adults. The person who takes primary responsibility for someone who cannot care fully for themselves is called the primary caregiver.

A recent personal study concerning elderly cancer patients caregivers show that most caregivers reported high or moderate levels of psychological distress, with an impact on their own health status.

In addition, family caregivers often report deficits in information about the disease, in training and skills related to their patients' care, and a lack of assistance from healthcare professionals.

The ability of the primary caregiver to meet the medical, material and emotional needs of the patient depends on their own resources (psychological, physical, intellectual, physical, financial) and on the diversity of their social network, but it also depends on the quality of the personalized support program (including information and training) that has been established for them.

Research hypotheses

Our hypothesis of research is that the needs and resources to help the couple " elderly patient/caregiver ", are at least in part socially determined and that the implementation of a personalized support plan to help the caregiver (PSP) taking into account needs, resources and expectations of the primary caregiver in addition to those of elderly patients with cancer may partly correct inequalities. The PSP should allow a better management of cancer, a lesser burden for the caregiver and a better quality of life for both the caregiver and the patient.

Intervention description

Prospective, interventional, randomized trial, with 118 patients in each group:

* an experimental interventional arm including an interview of the primary caregivers to identify their needs and expectations, the implementation of a "personalized support program", including telephone follow-up
* A control arm corresponding to the standard care. Caregiver aid is usually proposed when accompanying a sick relative in consultation or hospitalization.

All the "couples patient / caregiver' will benefit initially from:

1. a comprehensive geriatric assessment (elderly patients with cancer)
2. an assessment of caregiver burden by the Zarit burden interview (ZBI)
3. an assessment of subjective well-being
4. an individual assessment of the precariousness and health inequalities based on the score EPICES (Evaluation of precariousness and health inequalities in the health Centers)

Randomization will be stratified according to:

* living in the same household or not
* score of initial Zarit Burden Interview

Intervention Stage 1: A semi-structured interview centered on the caregiver's needs (COAT tool) Stage 2: guided questionnaires to assess the psychosocial situation of caregivers Stage 3: implementation of a multi-component PSP (information, counseling, listening time, training to help overcome their difficulties as a caregiver, planning for future care) Stage 4: at least one monthly phone interview Stage 5: 6 months follow up on the psychosocial characteristics of caregivers

Expected results in public health Our study will help to better define the way to take better account of the needs of the helper / helped couple, and reinforce the role of the coordinating nurse in the care pathways.

If our hypotheses can confirmed that there is a link between the caregivers needs and the social determinants of health and that the intervention has a positive impact on the caregivers burden and stress, it will suggest that this intervention not only acts favorably on social inequalities in health, but it can help reduce health care costs, as the caregiver exhaustion increases the risk of health expenditure (drug consumption, hospitalization of the patient and of the caregiver).

ELIGIBILITY:
Inclusion Criteria:

* Identification of a patient / caregiver couple
* Be the primary caregiver for at least one month of a subject

  * Age ≥70 years
  * With cancer
  * Who benefited a comprehensive geriatric assessement at University Lille Hospital or Centre Oscar Lambret
  * Affiliated to a social security or receiving an equivalent system of social protection
* caregiver able to understand the nature, purpose and methodology of the study
* caregiver able to cooperate in interviews and questionnaires
* Written informed consent of the caregiver and the cancer patient provided before any study specific procedures

Exclusion Criteria:

* Caregiver < 18 years old
* Legal inability or restricted legal ability
* Inability to attend or comply with interventions or follow-up scheduling, disability or difficulty preventing a proper understanding of trial instructions
* patient's life expectancy less than 6 months (clinical assessment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2014-12-11 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
change in caregiver burden (22 items Zarit Burden Interview) | 6 months

SECONDARY OUTCOMES:
Link between caregiver burden (ZBI) and the indicator of precariousness (EPICES score) | baseline evaluation
psychosocial characteristics of caregivers of patients with cancer | baseline and 6 months
  Caregiver Reaction Assessment (CRA) Carers' Assessment of Managing Index (CAMI) Inventory of social support (ISSB) Hospital Anxiety and Depression Scale (HADS) Cognitive Inventory of Subjective Distress (CISD) Subjective well-being scale (BES)
Link between caregiver burden and geriatric syndromes | baseline and 6 months
Link between caregiver burden and stage of cancer / time from cancer diagnosis | baseline
Match between caregiver personalized support plan (PSP) objectives and effective implemented PSP | 6 months
Time spent for the development and implementation of the caregiver personalized support plan | 6 months

OTHER OUTCOMES:
Relationship between needs and EPICES score | baseline

CONTACTS AND LOCATIONS:
Overall Officials: GAXATTE Cédric, MD, Study Chair — University Hospital, Lille
Locations (2):
- France (2):
  - Centre Oscar Lambret, Lille
  - University hospital, Lille, Lille

IPD SHARING:
Plan to Share IPD: Undecided